CLINICAL TRIAL: NCT03845452
Title: Retrospective Study : Muscle Mass or Muscle Function as a prédictive Tools for Outtcomme in Chronic Dialysis Patients
Brief Title: Muscle Mass or Muscle Function as a prédictive Tools for Outtcomme in Chronic Dialysis Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0447
Record Dates: First submitted 2019-02-18; First posted 2019-02-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2019-02

CONDITIONS: Chrnoic Haemodialysis Patients
Keywords: chronic kidney disease; muscle strength; muscle mass; lean body mass; physical activity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this study is to compare the association of muscle mass and functionality with mortality among chronic haemodialysis

* the involvement of malnutrition inflammation and atherogenesis syndrome (increase in C reactive protein and decrease in serum albumin) on voluntary muscle strength impairment and phyiscal activity.
* the relationship between voluntary muscle strength and mortality
* the relationship between voluntary muscle strength and physical activity

DETAILED DESCRIPTION:
Aim of this study is to compare the association of muscle mass and functionality with mortality among chronic haemodialysis

* the involvement of malnutrition inflammation and atherogenesis syndrome (increase in C reactive protein and decrease in serum albumin) on voluntary muscle strength impairment and phyiscal activity.
* the relationship between voluntary muscle strength and mortality
* the relationship between voluntary muscle strength and physical activity

ELIGIBILITY:
Inclusion criteria:

* chronic kidney disease patient with extrarenal replacement therapy by hemodialysis for at least 3 months
* stable clinical condition (absence of infection, stroke or acute decompensation)

Exclusion criteria:

* chronic kidney disease without extrarenal replacement therapy
* history of renal transplantation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chrnoic haemodialysis patients
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality at 2 years | 2 years
  Mortality at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul CRISTOL, Prof, Principal Investigator — CHU Lapeyronie, Department of Biochemistry and Hormonology, Montpellier, FRANCE
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Souweine JS, Pasquier G, Morena M, Patrier L, Rodriguez A, Raynal N, Ohresser I, Benomar R, Hayot M, Mercier J, Gouzi F, Cristol JP. Beyond sarcopenia: frailty in chronic haemodialysis patients. Clin Kidney J. 2024 Jun 29;17(7):sfae069. doi: 10.1093/ckj/sfae069. eCollection 2024 Jul. PMID 38983653